CLINICAL TRIAL: NCT04971694
Title: A Retrospective Chart Review Evaluating the Impact of Steroid, Diuretic, and Fluid Use Practice Trends in Extreme Premature Infants At Risk for Bronchopulmonary Dysplasia (BPD) At a Single Center Neonatal Intensive Care Unit
Brief Title: Impact of Steroid, Diuretic, and Fluid Use on BPD Outcomes
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Collaborators: Banner Health (Other); Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 830900795
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: BPD - Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Inclusion Group: Infants born at <30 weeks and/or <1500g that were admitted to BUMCP between January 1, 2019 and December 31, 2020
  Interventions: Other: No interventions or procedures

INTERVENTIONS:
Other: No interventions or procedures — This is a retrospective observational study and data will be collected from the subject's existing medical record. No interventions or procedures will be required for this study.

SUMMARY:
Assess the impact of steroid, diuretic, and fluid practices on BPD outcomes in extreme premature infants in the Banner - University Medical Center Phoenix (BUMCP) neonatal intensive care unit (NICU).

DETAILED DESCRIPTION:
The investigators propose performing a retrospective analysis of the current respiratory management methods to potentially find a correlation between the number of steroid doses administered, the timing of initiation of steroid therapy and the effect on premature infants at risk for developing BPD. The investigators are also going to explore the number and timing of diuretic medications and average fluid intake.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at <30 weeks and/or <1500g
* Admitted to BUMCP between January 1, 2019 and December 31, 2020

Exclusion Criteria:

* Infants that do not survive to 36 weeks CGA, when the determination of BPD is made
* Infants that are transferred to another hospital prior to 36 weeks CGA
* Out born infants
* Infants with life threatening congenital anomalies
* Investigator discretion as to other factors which might impact the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants admitted to the BUMCP NICU at <30 weeks and/or <1500 grams (g)
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2024-07-06 (Actual)

PRIMARY OUTCOMES:
To assess the impact of steroid practices on BPD outcomes in these infants | 30 days
  - The incidence of BPD stratified into three stages based on the type of support required at 36 weeks CGA
To assess the impact of steroid practices on BPD outcomes in these infants | 30 days
  - Presence of prenatal steroid administration
To assess the impact of steroid practices on BPD outcomes in these infants | 30 days
  - Administration of steroids to the infant

SECONDARY OUTCOMES:
To determine if steroid use has an impact on infant growth | 30 days
  - Collect growth and calculate the z-score at five intervals
To determine if steroid use has an impact on NICU length of stay (LOS) | 30 days
  - NICU LOS in days

OTHER OUTCOMES:
To determine if the average fluid intake in the first week of life influences the severity of BPD | 1-6 days
  - Fluid average from DOL 1-6
To determine if diuretic administration influences the severity of BPD | 1-6 days
  - If applicable, the DOL of first furosemide and/or chlorothiazide doses

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Valladolid, MD, Principal Investigator — Banner University Medical Center
Locations (1):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Northway WH Jr, Rosan RC, Porter DY. Pulmonary disease following respirator therapy of hyaline-membrane disease. Bronchopulmonary dysplasia. N Engl J Med. 1967 Feb 16;276(7):357-68. doi: 10.1056/NEJM196702162760701. No abstract available. PMID 5334613
- [Background] Guaman MC, Gien J, Baker CD, Zhang H, Austin ED, Collaco JM. Point Prevalence, Clinical Characteristics, and Treatment Variation for Infants with Severe Bronchopulmonary Dysplasia. Am J Perinatol. 2015 Aug;32(10):960-7. doi: 10.1055/s-0035-1547326. Epub 2015 Mar 4. PMID 25738785
- [Background] Jensen EA, Schmidt B. Epidemiology of bronchopulmonary dysplasia. Birth Defects Res A Clin Mol Teratol. 2014 Mar;100(3):145-57. doi: 10.1002/bdra.23235. Epub 2014 Mar 17. PMID 24639412
- [Background] Jensen EA, Dysart K, Gantz MG, McDonald S, Bamat NA, Keszler M, Kirpalani H, Laughon MM, Poindexter BB, Duncan AF, Yoder BA, Eichenwald EC, DeMauro SB. The Diagnosis of Bronchopulmonary Dysplasia in Very Preterm Infants. An Evidence-based Approach. Am J Respir Crit Care Med. 2019 Sep 15;200(6):751-759. doi: 10.1164/rccm.201812-2348OC. PMID 30995069
- [Background] Sward-Comunelli SL, Mabry SM, Truog WE, Thibeault DW. Airway muscle in preterm infants: changes during development. J Pediatr. 1997 Apr;130(4):570-6. doi: 10.1016/s0022-3476(97)70241-5. PMID 9108855
- [Background] Tiddens HA, Hofhuis W, Casotti V, Hop WC, Hulsmann AR, de Jongste JC. Airway dimensions in bronchopulmonary dysplasia: implications for airflow obstruction. Pediatr Pulmonol. 2008 Dec;43(12):1206-13. doi: 10.1002/ppul.20928. PMID 18991341
- [Background] O'Reilly M, Hooper SB, Allison BJ, Flecknoe SJ, Snibson K, Harding R, Sozo F. Persistent bronchiolar remodeling following brief ventilation of the very immature ovine lung. Am J Physiol Lung Cell Mol Physiol. 2009 Nov;297(5):L992-L1001. doi: 10.1152/ajplung.00099.2009. Epub 2009 Aug 28. PMID 19717553
- [Background] Ter Wolbeek M, Kavelaars A, de Vries WB, Tersteeg-Kamperman M, Veen S, Kornelisse RF, van Weissenbruch M, Baerts W, Liem KD, van Bel F, Heijnen CJ. Neonatal glucocorticoid treatment: long-term effects on the hypothalamus-pituitary-adrenal axis, immune system, and problem behavior in 14-17 year old adolescents. Brain Behav Immun. 2015 Mar;45:128-38. doi: 10.1016/j.bbi.2014.10.017. Epub 2014 Nov 8. PMID 25449580
- [Background] Cheong JL, Burnett AC, Lee KJ, Roberts G, Thompson DK, Wood SJ, Connelly A, Anderson PJ, Doyle LW; Victorian Infant Collaborative Study Group. Association between postnatal dexamethasone for treatment of bronchopulmonary dysplasia and brain volumes at adolescence in infants born very preterm. J Pediatr. 2014 Apr;164(4):737-743.e1. doi: 10.1016/j.jpeds.2013.10.083. Epub 2013 Dec 12. PMID 24332820
- [Background] Doyle LW, Cheong JL, Ehrenkranz RA, Halliday HL. Early (< 8 days) systemic postnatal corticosteroids for prevention of bronchopulmonary dysplasia in preterm infants. Cochrane Database Syst Rev. 2017 Oct 24;10(10):CD001146. doi: 10.1002/14651858.CD001146.pub5. PMID 29063585
- [Background] Zeng L, Tian J, Song F, Li W, Jiang L, Gui G, Zhang Y, Ge L, Shi J, Sun X, Mu D, Zhang L. Corticosteroids for the prevention of bronchopulmonary dysplasia in preterm infants: a network meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2018 Nov;103(6):F506-F511. doi: 10.1136/archdischild-2017-313759. Epub 2018 Feb 23. PMID 29475879
- [Background] Doyle LW, Cheong JL, Ehrenkranz RA, Halliday HL. Late (> 7 days) systemic postnatal corticosteroids for prevention of bronchopulmonary dysplasia in preterm infants. Cochrane Database Syst Rev. 2017 Oct 24;10(10):CD001145. doi: 10.1002/14651858.CD001145.pub4. PMID 29063594
- [Background] Onland W, De Jaegere AP, Offringa M, van Kaam AH. Effects of higher versus lower dexamethasone doses on pulmonary and neurodevelopmental sequelae in preterm infants at risk for chronic lung disease: a meta-analysis. Pediatrics. 2008 Jul;122(1):92-101. doi: 10.1542/peds.2007-2258. PMID 18595991
- [Background] Onland W, Offringa M, De Jaegere AP, van Kaam AH. Finding the optimal postnatal dexamethasone regimen for preterm infants at risk of bronchopulmonary dysplasia: a systematic review of placebo-controlled trials. Pediatrics. 2009 Jan;123(1):367-77. doi: 10.1542/peds.2008-0016. PMID 19117904
- [Background] Doyle LW, Ehrenkranz RA, Halliday HL. Postnatal hydrocortisone for preventing or treating bronchopulmonary dysplasia in preterm infants: a systematic review. Neonatology. 2010;98(2):111-7. doi: 10.1159/000279992. Epub 2010 Feb 12. PMID 20150750
- [Background] Peltoniemi OM, Lano A, Yliherva A, Kari MA, Hallman M; Neonatal Hydrocortisone Working Group. Randomised trial of early neonatal hydrocortisone demonstrates potential undesired effects on neurodevelopment at preschool age. Acta Paediatr. 2016 Feb;105(2):159-64. doi: 10.1111/apa.13074. Epub 2015 Nov 5. PMID 26058477
- [Background] Baud O, Maury L, Lebail F, Ramful D, El Moussawi F, Nicaise C, Zupan-Simunek V, Coursol A, Beuchee A, Bolot P, Andrini P, Mohamed D, Alberti C; PREMILOC trial study group. Effect of early low-dose hydrocortisone on survival without bronchopulmonary dysplasia in extremely preterm infants (PREMILOC): a double-blind, placebo-controlled, multicentre, randomised trial. Lancet. 2016 Apr 30;387(10030):1827-36. doi: 10.1016/S0140-6736(16)00202-6. Epub 2016 Feb 23. PMID 26916176
- [Background] Parikh NA, Kennedy KA, Lasky RE, McDavid GE, Tyson JE. Pilot randomized trial of hydrocortisone in ventilator-dependent extremely preterm infants: effects on regional brain volumes. J Pediatr. 2013 Apr;162(4):685-690.e1. doi: 10.1016/j.jpeds.2012.09.054. Epub 2012 Nov 8. PMID 23140612
- [Background] Parikh NA, Kennedy KA, Lasky RE, Tyson JE. Neurodevelopmental Outcomes of Extremely Preterm Infants Randomized to Stress Dose Hydrocortisone. PLoS One. 2015 Sep 16;10(9):e0137051. doi: 10.1371/journal.pone.0137051. eCollection 2015. PMID 26376074
- [Background] Kersbergen KJ, de Vries LS, van Kooij BJ, Isgum I, Rademaker KJ, van Bel F, Huppi PS, Dubois J, Groenendaal F, Benders MJ. Hydrocortisone treatment for bronchopulmonary dysplasia and brain volumes in preterm infants. J Pediatr. 2013 Sep;163(3):666-71.e1. doi: 10.1016/j.jpeds.2013.04.001. Epub 2013 May 21. PMID 23706359
- [Background] Oh W, Poindexter BB, Perritt R, Lemons JA, Bauer CR, Ehrenkranz RA, Stoll BJ, Poole K, Wright LL; Neonatal Research Network. Association between fluid intake and weight loss during the first ten days of life and risk of bronchopulmonary dysplasia in extremely low birth weight infants. J Pediatr. 2005 Dec;147(6):786-90. doi: 10.1016/j.jpeds.2005.06.039. PMID 16356432
- [Background] Slaughter JL, Stenger MR, Reagan PB. Variation in the use of diuretic therapy for infants with bronchopulmonary dysplasia. Pediatrics. 2013 Apr;131(4):716-23. doi: 10.1542/peds.2012-1835. Epub 2013 Mar 11. PMID 23478874
- [Background] Stewart A, Brion LP. Intravenous or enteral loop diuretics for preterm infants with (or developing) chronic lung disease. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD001453. doi: 10.1002/14651858.CD001453.pub2. PMID 21901676
- [Background] Stewart A, Brion LP, Ambrosio-Perez I. Diuretics acting on the distal renal tubule for preterm infants with (or developing) chronic lung disease. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD001817. doi: 10.1002/14651858.CD001817.pub2. PMID 21901679
- [Background] Sahni J, Phelps SJ. Nebulized furosemide in the treatment of bronchopulmonary dysplasia in preterm infants. J Pediatr Pharmacol Ther. 2011 Jan;16(1):14-22. PMID 22477820
- [Background] Segar JL. Neonatal diuretic therapy: furosemide, thiazides, and spironolactone. Clin Perinatol. 2012 Mar;39(1):209-20. doi: 10.1016/j.clp.2011.12.007. Epub 2011 Dec 29. PMID 22341547
- [Background] Demling RH, Will JA. The effect of furosemide on the pulmonary transvascular fluid filtration rate. Crit Care Med. 1978 Sep-Oct;6(5):317-9. doi: 10.1097/00003246-197809000-00003. PMID 569036
- [Background] Dikshit K, Vyden JK, Forrester JS, Chatterjee K, Prakash R, Swan HJ. Renal and extrarenal hemodynamic effects of furosemide in congestive heart failure after acute myocardial infarction. N Engl J Med. 1973 May 24;288(21):1087-90. doi: 10.1056/NEJM197305242882102. No abstract available. PMID 4697939
- [Background] Lundergan CF, Fitzpatrick TM, Rose JC, Ramwell PW, Kot PA. Effect of cyclooxygenase inhibition on the pulmonary vasodilator response to furosemide. J Pharmacol Exp Ther. 1988 Jul;246(1):102-6. PMID 3134540
- [Background] Almirall JJ, Dolman CS, Eidelman DH. Furosemide-induced bronchodilation in the rat bronchus: evidence of a role for prostaglandins. Lung. 1997;175(3):155-63. doi: 10.1007/pl00007563. PMID 9087943
- [Background] Greenberg RG, Gayam S, Savage D, Tong A, Gorham D, Sholomon A, Clark RH, Benjamin DK, Laughon M, Smith PB; Best Pharmaceuticals for Children Act-Pediatric Trials Network Steering Committee. Furosemide Exposure and Prevention of Bronchopulmonary Dysplasia in Premature Infants. J Pediatr. 2019 May;208:134-140.e2. doi: 10.1016/j.jpeds.2018.11.043. Epub 2018 Dec 20. PMID 30579586
- [Background] Hoffman DJ, Gerdes JS, Abbasi S. Pulmonary function and electrolyte balance following spironolactone treatment in preterm infants with chronic lung disease: a double-blind, placebo-controlled, randomized trial. J Perinatol. 2000 Jan-Feb;20(1):41-5. doi: 10.1038/sj.jp.7200307. PMID 10693099
- [Background] Bell EF, Acarregui MJ. Restricted versus liberal water intake for preventing morbidity and mortality in preterm infants. Cochrane Database Syst Rev. 2014;2014(12):CD000503. doi: 10.1002/14651858.CD000503.pub3. Epub 2014 Dec 4. PMID 25473815
- [Background] Kavvadia V, Greenough A, Dimitriou G, Forsling ML. Randomized trial of two levels of fluid input in the perinatal period--effect on fluid balance, electrolyte and metabolic disturbances in ventilated VLBW infants. Acta Paediatr. 2000 Feb;89(2):237-41. doi: 10.1080/080352500750028898. PMID 10709897
- [Background] Chou JH, Roumiantsev S, Singh R. PediTools Electronic Growth Chart Calculators: Applications in Clinical Care, Research, and Quality Improvement. J Med Internet Res. 2020 Jan 30;22(1):e16204. doi: 10.2196/16204. PMID 32012066
- [Background] Olaloko O, Mohammed R, Ojha U. Evaluating the use of corticosteroids in preventing and treating bronchopulmonary dysplasia in preterm neonates. Int J Gen Med. 2018 Jul 3;11:265-274. doi: 10.2147/IJGM.S158184. eCollection 2018. PMID 30013381